CLINICAL TRIAL: NCT00355329
Title: Randomized Control Trial of Using Tongue Acupuncture in Autistic Spectrum Disorder Using PET Scan for Clinical Correlation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PET-001
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Last update posted 2006-10-20 (Estimated); Status verified 1999-07

CONDITIONS: Autism; Autistic Disorder
Keywords: Traditional Chinese Medicine (TCM); Autism; Autistic Spectrum Disorder; Tongue Acupuncture (TAC); 18F-fluorodeoxyglucose Positron Emission Tomography (PET); children
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

INTERVENTIONS:
Procedure: Tongue Acupuncture (Procedure)

SUMMARY:
We aimed to use Tongue Acupuncture (TAC) to assess for any change in brain function.

DETAILED DESCRIPTION:
Autism or Autistic Spectrum Disorder is a neurodevelopmental disorder affecting language, communication, social interaction and behavior. Autism is a heterogeneous disorder makes the assessment of treatment difficult. Only few measures have been used in a standardized way to document the outcome of different modalities of treatment in autism. Most claims of treatment effect in autism have been quite anecdotal.

In Traditional Chinese acupuncture, nearly 400 acupoints on the body surface are interrelated to various functions. Acupuncture had been practiced in China for over 2 millennia. The surface acupoints are linked through 14 meridians to various organs or viscera of the human body. The approach in TCM, in sharp contrast to western medical concept, is a "holistic" approach with a more philosophical background of balancing the "Yin-and-Yang". The main objective of TCM is to improve health of body and mind.

The pathophysiological basis of TCM aimed to improve "energy" or "body-flow" ["de-qui" in Chinese]. Even a normal human subject will respond to acupuncture due to the flow of energy. The effect of acupuncture was hypothesized and proven in animal and human studies to be due to direct neural stimulation, changes in neurotransmitters such as endorphin, immunological markers and endocrinological signals. Thus, acupuncture is Thus, acupuncture is effective in chronic disorders, especially in neurological disorders.

We had demonstrated clinical efficacy of acupuncturing the surface or base of the tongue in specific acupoints in improving various functional modalities in patients with chronic neurological disorders such as cerebral palsy, stroke and drooling problems. In our experience, TCM approach for autism is more holistic. Autism is postulated as part of the spectrum of lower intelligence. Thus, the approach to autism is considered as lower intelligence due to "Heart-meridian and Kidney-meridian yin-yang imbalance" resulting in communication problem and "Liver-meridian yin-yang imbalance " leading to behavioral problems.

We attempted to use a different approach in looking at autism and to assess the efficacy of an innovative method in TCM in improving the functional status of these children. Specific acupoints in the tongue corresponding to various organs and meridians were used for autism. The organ and meridian concept in TCM model has been assumed as a fundamental basis to improve the behavior, cognition and communicative ability in children with autism. The objective is to study the efficacy of a short course of TAC in improving the overall functional status of autism.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of autism was made using standard criteria of the 4th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and Autism Diagnostic Interview-Revised (ADI-R).
* The diagnosis of autism was made if the score in the Childhood Autism Rating Scale (CARS)was greater than 30.

Exclusion Criteria:

* Children with associated neurological disorders such as Tuberous Sclerosis, Fragile X Syndrome and epilepsy.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30

PRIMARY OUTCOMES:
Autism Treatment Evaluation Checklist (ATEC) consisting of 4 subscales before (Week 0) and after (Week 8) acupuncture
Reynell Language Developmental Scale (RLDS) before (Week 0) and after (Week 8) acupuncture
Symbolic Play Test (SPT) before (Week 0) and after (Week 8) acupuncture
Functional Independence Measure for children (WeeFIM) with 3 domains before (Week 0) and after (Week 8) acupuncture
Clinical Global Impression Scale (CGIS) before (Week 0) and after (Week 8) acupuncture
18F-fluorodeoxyglucose Positron Emission Tomography (PET) before (Week 0) and after (Week 8) acupuncture

CONTACTS AND LOCATIONS:
Overall Officials: Wong Virginia, Principal Investigator — The University of Hong Kong
Locations (1):
- Duchess of Kent of Children Hospital, Hong Kong, Hong Kong